CLINICAL TRIAL: NCT05992766
Title: The Effect of Traditional Mat Exercises Versus Reformer Pilates and Hammock Yoga on Pain, Endurance, Balance, Disability, and Quality of Life in Individuals Who Had Chronic Back Pain
Brief Title: The Effect of Traditional Mat Exercises Versus Reformer Pilates and Hammock Yoga on Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Ass Prof, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/037
Record Dates: First submitted 2023-08-05; First posted 2023-08-15 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
Keywords: Chronic Back Pain; Reformer Pilates; Hammock Yoga; Physical Fitness; Quality of Life
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The participants were divided into 3 groups with closed envelope randomization method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reformer Pilates (Experimental): Reformer Pilates were performed, 2 days a week, for 4 weeks, in a total of 8 sessions (45 minutes each). The exercises of the Reformer Pilates were given as individual sessions by the physiotherapist. Reformer Exercises were explained by the physiotherapist in detail to understand the movement and starting position correctly, and the participants were then asked to perform the movements.
  Interventions: Other: Reformer Pilates
- Hammach Yoga (Experimental): Hammock Yoga were performed, 2 days a week, for 4 weeks, in a total of 8 sessions (45 minutes each). Hammock Yoga were given as individual sessions by the physiotherapist.
  Interventions: Other: Hammock Yoga
- Mat (Active Comparator): Traditional mat exercises were performed, 2 days a week, for 4 weeks, in a total of 8 sessions (45 minutes each). The mat exercises were applied as a home program. The exercises were visually given with detailed explanations on a piece of paper, and they were checked by telephone every week.
  Interventions: Other: Traditional mat exercises

INTERVENTIONS:
Other: Reformer Pilates — Reformer Pilates exercises activates the lumbopelvic muscles and supports functional movement. Activated muscles support the spine and reduce the load on the spine by correcting the posture, helping the core muscles such as the abdomen and spine stay healthier by attaching them to a neutral pelvis Pilates consists of a sliding platform working with the help of a pulley system specific to the use, allowing the individual to apply certain resistances, and providing the opportunity to exercise sitting, standing, or lying down.
  Arms: Reformer Pilates
Other: Hammock Yoga — Hammock Yoga is performed with a silk hammock, which is an auxiliary equipment. The most distinctive characteristic that makes Hammock Yoga different from other exercises is the spine traction provided by the upside-down posture, and the smooth and shiny silk hammock allows strengthening exercises. The Hammock Yoga aims to reduce the load on the spine by upside-down postures that defy the laws of physics.
  Arms: Hammach Yoga
Other: Traditional mat exercises — The mat exercises help build core strength, stamina, and motor control of the abdominal and lumbar trunk musculature. The exercises focus on the re-education of a precise co-contraction pattern of local muscles of the spine. Also mat exercise increases the level of endorphins and the stimulation of mechanoreceptors, causing biomechanical stress to support healing in tissues.
  Arms: Mat

SUMMARY:
The purpose of the present study was to examine the effects of traditional mat exercises, Reformer Pilates and Hammock Yoga approaches on pain, endurance, balance, disability, and quality of life of individuals who had Chronic Back Pain.

DETAILED DESCRIPTION:
Low back pain is among the leading musculoskeletal problems worldwide causing serious health expenditures. It can affect people of all ages in the community, but it is common in individuals between the fourth and fifth decades of life. Low back pain is divided into 3 subclasses according to the duration of the symptoms as Acute (lasting only a few weeks), Subacute (lasting about 6 to 12 weeks), and Chronic (lasting more than 12 weeks).Traditional exercise approaches are frequently used modalities in the treatment of Chronic Back Pain as an extremely valuable approach to preventing movement limitation, controlling existing pain, and regaining motor functions. Pilates exercises are very valuable for the treatment of low back pain because they provide stabilization. Pilates activates the lumbopelvic muscles and supports functional movement as an effective factor in reducing pain. Yoga is also a mind-body exercise discipline that includes both physical and mental aspects of pain with core strengthening, flexibility, relaxation, and breathing modalities.When the literature was reviewed, no study was detected examining the effectiveness of Hammock Yoga and Reformer Pilates in people who have Chronic Back Pain and compares it with traditional mat exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being within the 25-60 age range
* Having low back pain in the last 6 months .

Exclusion Criteria:

* The history of surgery in the lumbar region in the last 1 year,
* Diagnosed radiculopathy,
* Systemic diseases
* Malignancy,
* Performed regular physical activity,
* Using steroids and anti-inflammatory drugs in the physiotherapy program

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Pain characteristics | 4 weeks
  McGill Short Form was used at the beginning and end of the study to evaluate the qualitative characteristics of pain. The scale helps to learn about the sensory, emotional, and intensity component of pain. Fifteen items in the scale help define pain (11 sensory descriptors and 4 emotional descriptors). The participants were asked to rate their pain as 0=none, 1=less, 2=moderate, and 3=extreme, according to the intensity level. The total score was obtained by summing the scores given.
Disability | 4 weeks
  Disability (e.g., walking, sitting, standing, pain intensity, and sleeping) were evaluated with the Oswestry Disability Index, which consisted of 10 sections. A total score was obtained by scoring a Likert-type design ( 0-5 in each section). An increase in the score indicated an increased disability
Quality of Life | 4 weeks
  The World Health Organization Quality of Life-Bref (WHOQOL-Bref) Questionnaire was used to evaluate the quality of life. The questionnaire has 5 sections (Psychological Health, Physical Health, General Health, Social Relations, and Environmental Health).An increase in the score indicated an increased Quality of Life.
Pain intensity | 4 weeks
  A Visual Analog Scale was used to evaluate pain intensity. This scale is a straight horizontal line of fixed length, usually 100 mm. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Core Muscle Endurance Test | 4 weeks
  The forward plank test was used to measure the control and endurance of the back/core stabilizing muscles.The aim of this test was to hold an elevated position for as long as possible. Start with the upper body supported off the ground by the elbows and forearms, and the legs straight with the weight taken by the toes. The hip was lifted off the floor creating a straight line from head to toe. As soon as the subject was in the correct position, the stopwatch was started and time was recorded
Static Balance Test | 4 weeks
  The static balance was evaluated with single leg stance test. The participants were asked to pull their knees towards the abdomen and maintain this position while keeping their hands on their waists without disturbing the neutral pelvis (22). The time that passed until the position was broken was calculated and this test was repeated three times in total for both the right and left legs, and the maximum time was recorded in seconds.
Hip Muscle Endurance Test | 4 weeks
  The Single Leg Bridge Test was used to measure hip muscles endurance;The participants were asked to go to the bridge position with their supine hands-free at their sides and hips in the air, and while they were in this position, they were asked to keep the hip and knee flexion of the tested side and take the other leg into the air with the sole on the ground, and maintain the neutral position of the pelvis. When the test position was taken, the stopwatch was started and recorded the time until the participant broke the pelvis position.
Dynamic Balance Test | 4 weeks
  The dynamic balance was evaluated with the Star Excursion Balance Test. A total of 8 lines (anterolateral, anterior, anteromedial, medial, posteromedial, posterior, posterolateral, and lateral) of 1m length were drawn on a flat surface at 45 degree their centers converging. The individuals were then asked to reach the farthest point possible in each line with the tip of the other foot and the foot to be tested in the middle of the star. A resting period of 5 seconds was given after each stretch. If the balance was disturbed while reaching, the participants could not touch the lines, or gave full weight with their feet, the attempt was rejected and repeated. The distances that the individuals could reach and touch were recorded, and the test was repeated 3 times to record the maximum score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sorosky S, Stilp S, Akuthota V. Yoga and pilates in the management of low back pain. Curr Rev Musculoskelet Med. 2008 Mar;1(1):39-47. doi: 10.1007/s12178-007-9004-1. PMID 19468897
- [Background] Sherman KJ, Cherkin DC, Wellman RD, Cook AJ, Hawkes RJ, Delaney K, Deyo RA. A randomized trial comparing yoga, stretching, and a self-care book for chronic low back pain. Arch Intern Med. 2011 Dec 12;171(22):2019-26. doi: 10.1001/archinternmed.2011.524. Epub 2011 Oct 24. PMID 22025101
- [Background] Rydeard R, Leger A, Smith D. Pilates-based therapeutic exercise: effect on subjects with nonspecific chronic low back pain and functional disability: a randomized controlled trial. J Orthop Sports Phys Ther. 2006 Jul;36(7):472-84. doi: 10.2519/jospt.2006.2144. PMID 16881464
- [Background] Zhu F, Zhang M, Wang D, Hong Q, Zeng C, Chen W. Yoga compared to non-exercise or physical therapy exercise on pain, disability, and quality of life for patients with chronic low back pain: A systematic review and meta-analysis of randomized controlled trials. PLoS One. 2020 Sep 1;15(9):e0238544. doi: 10.1371/journal.pone.0238544. eCollection 2020. PMID 32870936
- [Background] Lim EC, Poh RL, Low AY, Wong WP. Effects of Pilates-based exercises on pain and disability in individuals with persistent nonspecific low back pain: a systematic review with meta-analysis. J Orthop Sports Phys Ther. 2011 Feb;41(2):70-80. doi: 10.2519/jospt.2011.3393. Epub 2010 Oct 22. PMID 20972339
- [Background] Pereira LM, Obara K, Dias JM, Menacho MO, Guariglia DA, Schiavoni D, Pereira HM, Cardoso JR. Comparing the Pilates method with no exercise or lumbar stabilization for pain and functionality in patients with chronic low back pain: systematic review and meta-analysis. Clin Rehabil. 2012 Jan;26(1):10-20. doi: 10.1177/0269215511411113. Epub 2011 Aug 19. PMID 21856719